CLINICAL TRIAL: NCT03294044
Title: The Effectiveness of Smart Health Management Program With Proactive Overcoming for Patients With Chronic Illness: Randomized Controlled Trial
Brief Title: The Effectiveness of Smart Health Management Program for Patients With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government); National Institute of Health, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Young Ho Yun, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HI16C0455-1
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Hypertension; Dyslipidemias; Diabetes Mellitus
Keywords: Self-Management IT Program
MeSH Terms: conditions — Hypertension; Dyslipidemias; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICT programs (Experimental): ICT programs that include health information learning by disease, and self-management based on Smart Management Strategy for Health (SMASH) are provided. After that, subjects will conduct self-management health care for 12 weeks. After 3 months, they finish self-management ICT programs, and then they fill out the questionnaire.
  Interventions: Behavioral: ICT programs
- A book about chronic disease (Active Comparator): Subjects in the group get a book about chronic disease for patients. After 3 months, they finish reading the materials, they fill out the questionnaire.
  Interventions: Behavioral: A book about chronic disease

INTERVENTIONS:
Behavioral: ICT programs — ICT programs that include health information learning by disease and self-management based on Smart Management Strategy for Health (SMASH).
  Arms: ICT programs
Behavioral: A book about chronic disease — A Take-home book about chronic disease are provided for self-education
  Arms: A book about chronic disease

SUMMARY:
This study verifies efficacy of Smart Health Management Program developed for patients with chronic illness. The aim of the study is to observe the changes in clinical indicators, quality of life and health related behaviors when providing self-management programs with ICT for chronic disease patients.

DETAILED DESCRIPTION:
This study is to demonstrate that chronic disease patients (hypertension, diabetes and dyslipidemia) with ICT-based self-management and educational program can improve clinical outcomes and overall health status, including quality of life and health habits.

In addition to the economic burden, people with chronic disease experience various psychosocial crises such as anxiety and depression, which causes the deterioration of overall quality of life and increases social burden. However, standard Chronic Care Model (CCM) have limitations in that they do not provide self-management strategies of the patient in detail. Therefore, to improve the effectiveness of the CCM model, it is required to propose a new approach to the utilization of IT-based self-management program that is currently being developed to increase accessibility and efficiency of health care service.

Primary outcomes of this study are as follow: Improvement of clinical indicators in patients with hypertension, diabetes and hyperlipidemia.

Participants in this study will respond a baseline questionnaire about health habits, health behavior patterns and quality of life, diet, exercise, etc. After that, participants will be allocated randomly into the intervention group and the control group. The intervention group will receive self-management and educational program with ICT ("S Healthing") while the control group will receive basic educational material with same contents on the disease. "S Healthing" is based ICT- program and includes educational contents and self-management program based on Smart Management Strategy for Health (SMASH). The intervention group will conduct self-management for 3 months through smart phone application and web program. Participants will receive a questionnaire about the quality of life and health habits with the clinical examination 3 months after baseline survey was conducted. The result from two questionnaires (baseline, post-intervention) and clinical outcomes will be compiled and be compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Subject 19 years old and more
* Subject who understands the purpose of the study and signs with informed consent form
* Subject with chronic disease (hypertension, diabetes, dyslipidemia)
* Subject with more than one Poor Disease Control Indicator

  1. HbA1C 7.0% or more
  2. Systolic BP 140mmHg or more
  3. LDL-cholesterol 130mg/dL or more
* Subjects who use smart phones and PCs (those who can use ICT-based health care programs)

Exclusion Criteria:

* Inability to speak, understand, or write Korean
* Inability to understand the contents of the provided materials due to poor eyesight and hearing
* Medical conditions that would limit adherence to participation of the clinical trial (as confirmed by their referring physician; e.g. dyspnea, severe depression and other mental disorders)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Success in clinical outcomes of Hypertension from baseline to 3 months | Baseline, 3 months post-intervention
  Change in Systolic blood pressure(mmHg)
Success in clinical outcomes of Dyslipidemia from baseline to 3 months | Baseline, 3 months post-intervention
  Change in LDL Cholesterol (mg/dL)
Success in clinical outcomes of primary disease Diabetes from baseline to 3 months | Baseline, 3 months post-intervention
  Change in HbA1c (%)

SECONDARY OUTCOMES:
Health behavior patterns | Baseline, 3 months post-intervention
  We identify health habits by dividing into five steps according to the TTM stage. We evaluate increase in maintenance rate of health behavior patterns.
Depression | Baseline, 3 months post-intervention
  Change in depression score (PHQ-9)
Health Management Strategies | Baseline, 3 months post-intervention
  We use Smart Management Strategy for Health Assessment Tool (SAT) to assess their self-management (SM) strategies of health by themselves. We evaluate improvement of Health Management Strategies.
Quality of life (SF-12) | Baseline, 3 months post-intervention
  Improvement of quality of life (SF-12)
Quality of life (Mcgill QOL) | Baseline, 3 months post-intervention
  Improvement of quality of life (Mcgill QOL)
Quality of life (Euro-QoL) | Baseline, 3 months post-intervention
  Improvement of quality of life (Euro-QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University, Seoul, South Korea

REFERENCES:
- [Derived] Yun YH, Kang E, Cho YM, Park SM, Kim YJ, Lee HY, Kim KH, Lee K, Koo HY, Kim S, Rhee Y, Lee J, Min JH, Sim JA. Efficacy of an Electronic Health Management Program for Patients With Cardiovascular Risk: Randomized Controlled Trial. J Med Internet Res. 2020 Jan 22;22(1):e15057. doi: 10.2196/15057. PMID 32012053